CLINICAL TRIAL: NCT06577077
Title: Randomized Clinical Trial to Evaluate the Efficacy and Safety of Product CM9241GRU in Relieving Nasal Symptoms in Perennial Allergic Rhinitis
Brief Title: Efficacy/ Safety of Product CM9241GRU in Patients With Perennial Allergic Rhinitis
Acronym: RESPIRE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH-DCG-03(03/21)
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product CM9241GRU (Experimental)
  Interventions: Drug: Product CM9241GRU
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Product CM9241GRU — 01 tablet in the morning and 01 tablet in the evening for 14 days
  Arms: Product CM9241GRU
Drug: Placebo — 01 tablet in the morning and 01 tablet in the evening for 14 days
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of CM9241GRU versus placebo in the treatment of perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes aged 18 and over
* Ability to understand and consent to participate in this clinical research, expressed by signing the Informed Consent Form (ICF)
* Participants with a diagnosis of perennial allergic rhinitis, as determined by a history of symptoms related to non-seasonal allergen exposure for at least 9 months in the 12 months prior to the screening visit.

Exclusion Criteria:

* Participants who have had nasal surgery in the six (6) months prior to the screening visit, or who have obvious external structural abnormalities that interfere with nasal airflow and are considered clinically relevant by the investigator;
* Participants with non-allergic rhinitis (e.g. vasomotor, infectious, medication or drug-induced rhinitis) or seasonal allergic rhinitis;
* Participants with a current diagnosis or history of chronic rhinosinusitis, chronic purulent postnasal drip in the two (2) years prior to the screening visit;
* Participants diagnosed with asthma requiring regular use of systemic or inhaled corticosteroids; uncontrolled asthma (ACT: 5-15); partially controlled asthma (ACT: 16-19);
* Participants with a history of immunotherapy treatment in the 2 years prior to the screening visit;
* Participants with an upper respiratory tract infection or rhinosinusitis requiring antibiotic treatment in the 14 days prior to the screening visit and the randomization visit;
* Participants with an upper respiratory tract viral infection in the 7 days prior to the screening and randomization visits;
* Participants with severe hypertension, severe coronary artery disease, arrhythmias, glaucoma, hyperthyroidism, prostatic hypertrophy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Absolute reduction in the evening reflective total nasal symptom score (rTNSS) | 14 days
  Absolute reduction in the evening reflective total nasal symptom score (rTNSS) evaluated 14 days after starting treatment compared to the baseline evening rTNSS.

IPD SHARING:
Plan to Share IPD: No